CLINICAL TRIAL: NCT07339280
Title: "The Effect of Probiotics on the Degree of Dyspnea, Lung Function, and Inflammatory Mediators in Patients With Chronic Obstructive Pulmonary Disease (COPD)."
Brief Title: Probiotics in COPD: Effects on Symptoms, Lung Function, and Inflammation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Split (Other)
Collaborators: Abela Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Andrea Anić Matić,MD, Principal Investigator, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHS-COPD-PROBIO-2025; 2181-147/01-06/LJ.Z.-25-02 (Registry Identifier: Ethics Committee of University Hospital Split)
Record Dates: First submitted 2026-01-02; First posted 2026-01-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: COPD; COPD (Chronic Obstructive Pulmonary Disease); Probiotic; Probiotic Supplement
Keywords: COPD; Chronic Obstructive Pulmonary disease; mMRC; dyspnea; CAT; Interleukin-6; Probiotics; probiotic supplement; dietary supplement
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Probiotics; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Double-blinded
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic arm (Active Comparator): Participants will receive two capsules once daily of a probiotic dietary supplement for 16 weeks. The product will be coded to ensure blinding.
  Interventions: Dietary Supplement: Probiotic Capsule
- Placebo arm (Placebo Comparator): Participants will receive two capsules once daily of a placebo preparation for 16 weeks. The product will be coded to ensure blinding.
  Interventions: Dietary Supplement: placebo capsule

INTERVENTIONS:
Dietary Supplement: Probiotic Capsule — The participants will take two probiotic capsules per day for 16 weeks, containing S. boulardii, Lactobacillus plantarum LP 6596, and Lactobacillus plantarum HEAL9. The product will be coded for blinding purposes.
  Other Names: Lactobacillus plantarum; Lac.plantarum HEAL9; Lac.plantarum LP 6596; Saccharomyces boulardii; dietary supplement; probiotic supplement
  Arms: Probiotic arm
Dietary Supplement: placebo capsule — Participants will receive two capsules per day for 16 weeks, a placebo preparation that is identical in composition and form to the probiotic but does not contain an active substance. The product will be coded for blinding purposes.
  Other Names: placebo; placebo control
  Arms: Placebo arm

SUMMARY:
The goal of this randomized, placebo controlled, double-blind clinical trial is to find out whether a probiotic supplement can help adults with chronic obstructive pulmonary disease (COPD) breathe better and better control their symptoms. The study will try to answer does taking a probiotic supplement, compare with a placebo, reduce shortness of breath, does it improve daily COPD symptoms or change stool patterns by using validated questionnaires; does it affect lung function or inflammation. The results of this study may contribute to a better understanding of the disease, the application of new therapeutic options, and provide a foundation for future research.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a progressive respiratory condition characterized by persistent symptoms such as shortness of breath, chronic cough, sputum production, and periods of acute worsening. It is also associated with ongoing systemic inflammation, which contributes to symptom severity, impaired lung function, and increased risk of exacerbations. Emerging evidence suggests that the gut-lung axis may play a significant role in this inflammatory process. Probiotics, which help restore a healthy microbial balance and support gut barrier integrity, have been proposed as a potential strategy to modulate inflammation and respiratory symptoms. Several studies have suggested that probiotics may reduce respiratory symptoms, improve lung function and lower systemic inflammation in people with COPD.

This randomized study is designed to evaluate whether a probiotic supplement (Saccharomyces boulardii, Lactobacillus plantarum LP 6596, and Lactobacillus plantarum HEAL9) can improve shortness of breath, overall symptom burden, lung function, and selected inflammatory markers in adults with stable COPD compared with placebo. Participants will be recruited from multiple clinical centers and will continue their usual COPD therapy throughout the study period. A total of 60 adult participants with a confirmed diagnosis of COPD, stable disease and baseline dyspnea of mMRC (modified Medical Research Council) ≥ 1 will be randomized to receive either a probiotic supplement or placebo for 16 weeks. They will take either the probiotic supplement or placebo 2 capsules once daily for 16 weeks and will be examined at three clinic visits for symptom questionnaires- mMRC scale of dyspnea, CAT (COPD Assessment Test) and Bristol Stool Scale, blood sampling, and spirometry testing. Between clinic visits, participants will have regular telephone checks every 4 weeks to assess symptoms, adherence to the study product and possible side effects.

This trial aims to provide a more comprehensive understanding of how probiotic supplementation may influence dyspnea, quality of life, inflammatory activity, and respiratory function in COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a previously established diagnosis of COPD, regardless of the degree of airflow obstruction on pulmonary function testing.
2. Age over 18 years, regardless of sex.
3. Stable disease without exacerbations during the past two months (8 weeks).
4. Stable disease without changes to maintenance therapy during the past two months (8 weeks).
5. Patients with an mMRC score of 1 or higher.
6. Signed informed consent.

Exclusion Criteria:

1. patients diagnosed with serious comorbidities such as severe cardiovascular diseases (severe heart failure, acute coronary syndrome, or percutaneous coronary intervention within 6 months, uncontrolled tachy/bradyarrhythmias), patients with severe renal failure and a placed central venous catheter, patients with severe liver damage (Child-Pugh class C), patients with infectious hepatitis or HIV, active bloody diarrhea;
2. patients undergoing active oncological and hematological treatment;
3. patients who have had a stroke within the past 3 months;
4. transplanted patients, including allograft recipients;
5. patients on long-term systemic corticosteroid and immunosuppressive therapy (oral or intravenous form) as well as antifungal therapy,
6. patients who have had a COPD exacerbation within the past two months and are not in a stable condition,
7. patients diagnosed with asthma,
8. patients with a history of lung surgery or serious respiratory diseases other than COPD (active tuberculosis, sarcoidosis, pulmonary fibrosis, severe bronchiectasis, pulmonary aspergillosis, etc.),
9. patients who have recently participated in other clinical trials or have received experimental therapy,
10. patients with a history of severe allergic reactions or hypersensitivity to the components of the probiotic preparation,
11. patients with active alcoholism or drug addiction,
12. patients with severe psychiatric diagnoses or those with significant physical or cognitive limitations that would interfere with following the study protocol,
13. patients who have recently undergone surgery,
14. pregnant or breastfeeding women,
15. patients who have taken any probiotic preparations within one month before the start of the study,
16. patients whose COPD treatment is changed during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
mMRC scale of dyspnea | 8 weeks
  The primary objective of this study is to assess the degree of change in dyspnea, measured using the validated mMRC (Modified Medical Research Council) questionnaire in patients with COPD eight weeks after administration of the probiotic dietary supplement.

SECONDARY OUTCOMES:
CAT questionnaire | 8, 16 weeks
  To evaluate the effect of probiotic therapy on symptom control and quality of life in COPD patients using the validated CAT (COPD Assessment Test) questionnaire after 4, 8, 12, and 16 weeks of probiotic administration.
Bristol stool scale | 8, 16 weeks
  To assess the effect of probiotic therapy on stool appearance using the Bristol Stool Scale at baseline and after 8 and 16 weeks of probiotic administration.
mMRC | 4,12,16 weeks
  To evaluate changes in dyspnea severity on the mMRC scale after 4, 12, and 16 weeks of probiotic administration.
IL-6 | 8 weeks
  Changes in laboratory-measured IL-6 (interleukin-6) levels at baseline and after 8 weeks of probiotic administration.
Complete blood count | 8 and 16 weeks
  To investigate the effect of probiotics on changes in concentration of total leukocyte count (×10⁹/L) with differential ((concentration of neutrophil count (×10⁹/L) , eosinophil count (×10⁹/L), monocyte (×10⁹/L) and lymphocyte count (×10⁹/L)) at baseline and after 8 and 16 weeks.
Fibrinogen | 8 and 16 weeks
  To evaluate changes in serum concentration of fibrinogen (g/L) from baseline and after 8 and 16 weeks of probiotic administration.
CRP | 8 and 16 weeks
  To evaluate changes in serum concentration of CRP (C-reactive protein) in mg/L from baseline and after 8 and 16 weeks of probiotic administration.
Metabolic blood parameters-glucose | 8, 16 weeks
  To assess changes in concentration of plasma glucose (mmol/L) measured at baseline and after 8 and 16 weeks of probiotic administration.
Metabolic blood parameters-urea | 8, 16 weeks
  To assess changes in urea concentration (mmol/L) measured at baseline, 8 weeks, and 16 weeks of probiotic administration.
Metabolic blood parameters-creatinine | 8, 16 weeks
  To assess changes in creatinine concentration (µmol/L) measured at baseline, 8 weeks, and 16 weeks.
Metabolic blood parameters-liver enzymes | 8, 16 weeks
  To assess changes in activity of Aspartate Aminotransferase (AST) A (U/L), Alanine Aminotransferase (ALT) (U/L) and Gamma-Glutamyl Transferase (GGT) (U/L) at baseline and after 8 and 16 weeks of probiotic administration.
Metabolic blood parameters-electrolytes | 8, 16 weeks
  To assess changes in concentration of sodium (mmol/L), potassium (mmol/L), and chloride (mmol/L) at baseline, after 8 and 16 weeks of probiotic administration.
Metabolic blood parameters-lipid profile | 8, 16 weeks
  To assess changes in concentration of total cholesterol (mmol/L), High-Density Lipoprotein-HDL(mmol/L), Low-Density Lipoprotein-LDL(mmol/L), triglycerides (mmol/L) at baseline, 8 weeks, and 16 weeks of probiotic administration.
Lung function | 16 weeks
  To evaluate the effect of probiotics on spirometry-derived values: FEV₁% (forced expiratory volume in one second) (L), FVC% (forced vital capacity) (L), and the FEV₁/FVC ratio after bronchodilator testing at baseline and after 16 weeks of probiotic administration .
Acute exacerbations | 16 weeks
  To investigate the effect of probiotic strains on the incidence of acute exacerbations after 16 weeks.
Correlation IL-6 and CRP | 8 weeks
  To determine the correlation between IL-6 concentration and CRP after 8 weeks of probiotic administration.
Other correlations | 16 weeks
  To determine the correlation between CRP concentration and spirometry findings (FEV₁ and the FEV₁/FVC ratio); correlation between fibrinogen levels and spirometry findings (FEV₁ and the FEV₁/FVC ratio); correlation between leukocyte count and spirometry findings (FEV₁ and the FEV₁/FVC ratio) after 16 weeks of probiotic administration.
BMI | 16 weeks
  To evaluate the effect of probiotic strain administration on changes in body mass index (BMI) after 16 weeks of probiotic administration.

CONTACTS AND LOCATIONS:
Locations (5):
- Croatia (5):
  - General Hospital Karlovac, Karlovac
  - University Hospital Split, Split
  - General Hospital Sibenik, Šibenik
  - General Hospital Vinkovci, Vinkovci
  - University Hospital Centre Sestre milosrdnice, Zagreb

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves sensitive health information, and data sharing is not covered by the informed consent form or approved by the ethics committee. Only aggregated, anonymized study results will be made publicly available.

REFERENCES:
- [Background] Koblizek V, Milenkovic B, Barczyk A, Tkacova R, Somfay A, Zykov K, Tudoric N, Kostov K, Zbozinkova Z, Svancara J, Sorli J, Krams A, Miravitlles M, Valipour A. Phenotypes of COPD patients with a smoking history in Central and Eastern Europe: the POPE Study. Eur Respir J. 2017 May 11;49(5):1601446. doi: 10.1183/13993003.01446-2016. Print 2017 May. PMID 28495687
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Karim A, Muhammad T, Shahid Iqbal M, Qaisar R. A multistrain probiotic improves handgrip strength and functional capacity in patients with COPD: A randomized controlled trial. Arch Gerontol Geriatr. 2022 Sep-Oct;102:104721. doi: 10.1016/j.archger.2022.104721. Epub 2022 May 10. PMID 35567889
- [Background] Su Z, Ma C, Ru X, Zhang S, Wu C, Huang Y, Cen H, Yin Z, Zhang J. Effects of probiotic treatment on patients and animals with chronic obstructive pulmonary disease: a systematic review and meta-analysis of randomized control trials. Front Cell Infect Microbiol. 2024 Sep 11;14:1411222. doi: 10.3389/fcimb.2024.1411222. eCollection 2024. PMID 39324058
- [Background] Patibandla S, Bhatt N, Lief S, Beauti SM, Ansari AZ. Gut Microbiota Modulation in the Management of Chronic Obstructive Pulmonary Disease: A Literature Review. Cureus. 2024 Aug 14;16(8):e66875. doi: 10.7759/cureus.66875. eCollection 2024 Aug. PMID 39280360
- [Background] Panahi Y, Ghanei M, Vahedi E, Mousavi SH, Imani S, Sahebkar A. Efficacy of probiotic supplementation on quality of life and pulmonary symptoms due to sulfur mustard exposure: a randomized double-blind placebo-controlled trial. Drug Chem Toxicol. 2017 Jan;40(1):24-29. doi: 10.3109/01480545.2016.1166250. Epub 2016 Apr 14. PMID 27079636
- [Background] Aghamohammadi M, Ghodrati S, Jalili N, Jafari R, Rafiee E, Kamali K, Ghasemi M, Alizargar J. Effects of the oral probiotic Familact on dyspnea management in COPD patients: A randomized controlled trial. Heart Lung. 2025 May-Jun;71:63-68. doi: 10.1016/j.hrtlng.2025.02.002. Epub 2025 Feb 27. PMID 40020522
- [Background] Ertan Yazar E, Niksarlioglu EY, Yigitbas B, Bayraktaroglu M. How to Utilize CAT and mMRC Scores to Assess Symptom Status of Patients with COPD in Clinical Practice? Medeni Med J. 2022 Jun 23;37(2):173-179. doi: 10.4274/MMJ.galenos.2022.06787. PMID 35735170
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Nishimura K, Izumi T, Tsukino M, Oga T. Dyspnea is a better predictor of 5-year survival than airway obstruction in patients with COPD. Chest. 2002 May;121(5):1434-40. doi: 10.1378/chest.121.5.1434. PMID 12006425
- [Background] Sethi DK, Rhodes J, Ferris R, Banka R, Clarke A, Mishra EK. Breathlessness Predicts Mortality in Adults: A Systematic Review and Meta-Analysis. Cureus. 2023 May 18;15(5):e39192. doi: 10.7759/cureus.39192. eCollection 2023 May. PMID 37332470
- [Background] Kantatong T, Deesomchok A, Panpanich R, Sungkarat S, Siviroj P. Predicting quality of life in chronic obstructive pulmonary disease patients living in the rural area of chiang mai province, thailand. TOPHJ [Internet]. 2020 July 30 [cited 2025 Nov 1];13(1):357-64. Available from: https://openpublichealthjournal.com/VOLUME/13/PAGE/357/
- [Background] Agusti A, Celli BR, Criner GJ, Halpin D, Anzueto A, Barnes P, Bourbeau J, Han MK, Martinez FJ, Montes de Oca M, Mortimer K, Papi A, Pavord I, Roche N, Salvi S, Sin DD, Singh D, Stockley R, Lopez Varela MV, Wedzicha JA, Vogelmeier CF. Global Initiative for Chronic Obstructive Lung Disease 2023 Report: GOLD Executive Summary. Am J Respir Crit Care Med. 2023 Apr 1;207(7):819-837. doi: 10.1164/rccm.202301-0106PP. No abstract available. PMID 36856433
- [Background] MDCalc [Internet]. [cited 2025 Oct 7]. Mmrc (Modified medical research council) dyspnea scale. Available from: https://www.mdcalc.com/calc/4006/mmrc-modified-medical-research-council-dyspnea-scale
- [Background] Huang H, Huang X, Zeng K, Deng F, Lin C, Huang W. Interleukin-6 is a Strong Predictor of the Frequency of COPD Exacerbation Within 1 Year. Int J Chron Obstruct Pulmon Dis. 2021 Oct 28;16:2945-2951. doi: 10.2147/COPD.S332505. eCollection 2021. PMID 34737559
- [Background] Li CL, Liu SF. Exploring Molecular Mechanisms and Biomarkers in COPD: An Overview of Current Advancements and Perspectives. Int J Mol Sci. 2024 Jul 4;25(13):7347. doi: 10.3390/ijms25137347. PMID 39000454
- [Background] Global Initiative for Chronic Obstructive Lung Disease - GOLD [Internet]. [cited 2025 Oct 7]. Global initiative for chronic obstructive lung disease. Available from: https://goldcopd.org/
- [Background] Research randomizer [Internet]. [cited 2025 Oct 7]. Available from: https://www.randomizer.org/.